CLINICAL TRIAL: NCT01141621
Title: The Dallas Hereditary Spherocytosis Cohort Study
Status: Terminated | Type: Observational
Why Stopped: Insufficient staff to continue pursuing project
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IRB # 022010-024
Record Dates: First submitted 2010-06-04; First posted 2010-06-10 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Hereditary Spherocytosis
Keywords: HS; congenital hemolytic anemia; splenectomy; quality of life
MeSH Terms: conditions — Spherocytosis, Hereditary; Anemia, Hemolytic, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to

1. better characterize the short term and long term natural history of hereditary spherocytosis (HS) including diagnosis, complications, and indications for and response to splenectomy
2. evaluate and describe the health-related quality of life in children with HS.

DETAILED DESCRIPTION:
Patients with a new or established diagnosis of HS seen at Children's Medical Center will be asked to enroll in the study. Previous and current medical records will be reviewed to systematically catalogue their history of HS, including diagnosis, complications, hospitalizations, medications and laboratory data. Health-related quality of life questionnaires will be given to the patients and their parents at enrollment and periodically during the follow-up. Those who agree will have up to three small samples of blood collected and frozen for future laboratory studies of complications associated with HS and/or splenectomy.

We anticipate enrolling approximately 200 children and young adults with HS in this study and following them until adulthood (age 18-21 years).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS with or without prior splenectomy
* Age 0 - 21 years
* Spanish-speaking subjects are eligible to participate

Exclusion Criteria:

* Unable to provide contact information for follow-up

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Center for Cancer and Blood Disorders outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | Approximately at 5 years
  PedsQL measurement

SECONDARY OUTCOMES:
Primary indications for splenectomy | Approximately at 5 years
  Primary indication for splenectomy determined at time of splenectomy, if performed.
Complications of HS | Approximately at 5 years and at 10 years
Complications of splenectomy | Approximately at 5 years
Diagnosis of HS | At enrollment